CLINICAL TRIAL: NCT02345720
Title: Effects on Ocular Tissues of Vistakon® Investigational Multifocal Contact Lenses - Asian Population Study
Brief Title: Effects of Multifocal Contact Lens on Ocular Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CR-5632
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Results first posted 2016-10-05 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2016-10

CONDITIONS: Visual Acuity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- etafilcon - PVP (multi-focal) (Experimental): The investigational soft contact lenses will be worn in a daily wear modality for 30 days over the course of the study.
  Interventions: Device: etafilcon - PVP (multi-focal)

INTERVENTIONS:
Device: etafilcon - PVP (multi-focal) — The investigational contact lens must be worn at least six hours daily.

SUMMARY:
The purpose of this study is to evaluate the etafilcon - PVP (multi-focal)

ELIGIBILITY:
Inclusion Criteria:

1. The subject must read, understand, and sign the statement of Informed Consent and receive a fully executed copy of the form.
2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. The subject must be between 40 and 70 years of age.
4. The subject's vertex corrected spherical equivalent distance refraction must be in the range of 1.00 too -5.75 in each eye.
5. The subject must identify themselves as Asian by self-report and have eyes and eyelids with an automatically Asian appearance.
6. The subject's refractive cylinder must be less than or equal to -0.75D in each eye.
7. The subject's ADD power must be in the range of +0.75 D to +2.5 D in each eye.
8. The subject must have best corrected visual acuity of 20/20-3 or better in each eye.
9. Subjects own a wearable pair of spectacles, if required for their distance vision.
10. The subject must be an adapted soft contact lens wearer in both eyes (i.e. worn lenses a minimum of 5 days per week for at least 8 hours per day, for one month or more duration).
11. The subject must already be wearing a presbyopic contact lens correction (e.g. reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire".

Exclusion Criteria:

1. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued)
2. Any ocular or systemic allergies that contraindicate contact lens wear.
3. Any ocular or systemic disease, autoimmune disease, or use of medication, that will contraindicate contact lens wear.
4. Any ocular abnormality that may interfere with contact lens wear.
5. Use of any ocular medications, with the exception of rewetting drops.
6. Any previous intraocular surgery (e.g. radial keratotomy, PRK, LASIK, etc.).
7. Any grade 3 or greater slit lamp findings (e.g. edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) which may contraindicate contact lens wear.
8. History of herpetic keratitis.
9. Any ocular infection or inflammation.
10. Any corneal distortion or irregular cornea.
11. History of binocular vision abnormality or strabismus.
12. Any infectious disease (e.g. hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g. HIV).
13. History of diabetes.
14. Habitual wearer of etafilcon-A contact lens material.
15. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 23 subjects were enrolled in this study. Of the enrolled subjects, 3 did not meet the eligibility criteria and 20 were dispensed a study lens. All dispensed subjects completed the study.
Groups:
- Etafilcon PVP (Multi-focal): All subjects wore the same study lenses throughout the duration of this study.
Period: Overall Study
Arm/Group | Etafilcon PVP (Multi-focal)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All subjects that were dispensed a study lens.
Arm/Group | Etafilcon PVP (Multi-focal)
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.6 (6.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 5
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 20
Region of Enrollment [Number; unit: Participants]
  United Kingdom | 20

OUTCOME MEASURES:

1. Primary Outcome: Upper Eye Lid Margin Staining
Description: Upper Eye Lid Margin Staining is assessed via Ocular Photography using proprietary algorithm. The average grade across upper eye lid margin was reported in mm^2.
Time Frame: 30 days Post wear
Population: The analysis population consists of all subjects that were dispensed a study lens.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Etafilcon PVP (Multi-focal)
Number analyzed (Participants) | 20
mm^2 | 1.96 (1.03)

2. Primary Outcome: Limbal Staining
Description: Measured via Ocular Photography using proprietary algorithm. The limbal conjunctival lissamine green staining average surface area in % of the overall limbal area was reported.
Time Frame: 30 Days Post Wear
Population: The analysis population consist of all subjects that were dispensed a study lens.
Measure: Mean (Standard Deviation); unit: percentage of limbal area
Arm/Group | Etafilcon PVP (Multi-focal)
Number analyzed (Participants) | 20
percentage of limbal area
  Nasal | 1.03 (1.30)
  Temporal | 0.68 (1.38)

3. Primary Outcome: Corneal Staining
Description: The corneal fluorescein staining average surface area in % of the upper corneal quadrant was reported.
Time Frame: 30 Days Post Wear
Population: The analysis population consists of all subjects that were dispensed a study lens.
Measure: Mean (Standard Deviation); unit: percentage of upper corneal quadrant
Arm/Group | Etafilcon PVP (Multi-focal)
Number analyzed (Participants) | 20
percentage of upper corneal quadrant | 0.05 (0.12)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 3 months.
Arm/Group | Etafilcon PVP (Multi-focal)
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days